CLINICAL TRIAL: NCT02033200
Title: A Double-Blind, Randomized, Placebo-Controlled, Single-Dose, Parallel Study to Assess the Effects of Avanafil (STENDRA™) on Multiple Parameters of Vision, Including, But Not Limited to Visual Acuity, Intraocular Pressure, Pupillometry, and Color Vision Discrimination, in Healthy Male Subjects
Brief Title: Safety Study Looking at the Effects of Stendra on Vision
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TA-402
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Vision
Keywords: vision; Stendra; avanafil; PDE5 inhibitor; visual acuity; intraocular pressure; pupillometry; color vision discrimination; healthy males
MeSH Terms: interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Stendra 200 mg
  Interventions: Drug: Stendra 200 mg; Drug: Placebo
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Stendra 200 mg; Drug: Placebo

INTERVENTIONS:
Drug: Stendra 200 mg
  Other Names: avanafil
Drug: Placebo

SUMMARY:
The purpose of this study is to see if Stendra causes any changes in vision, eye pressure, pupil dilation, and color vision in healthy males.

DETAILED DESCRIPTION:
The objectives of this study are to assess the effect of Stendra on visual acuity, intraocular pressure, pupillometry, and color vision discrimination in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males 18 to 45 years of age, inclusive
* Non-tobacco user for at least 6 months prior to first dose

Exclusion Criteria:

* History or presence of retinal disease or any vision defects including color vision
* Intraocular pressure value ≥ 22mm Hg
* Resting heart rate < 45 or > 90 beats per minute (3 rechecks)
* Systolic blood pressure < 90 or > 140 mm Hg or Diastolic blood pressure < 50 or >90 mm Hg (3 rechecks)
* Initiation or change in dose of any α-blockers 14 days prior to randomization

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion Inc, Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: healthy male adults between the ages of 18 and 45
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (7.67) | 35.1 (7.67) | 35.0 (7.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 34 | 66
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 33 | 35 | 68
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Color Vision Discrimination 1 Hour Post Dosing
Description: Color vision discrimination was performed using the Lanthony 40-Hue Test according to Farnsworth-Munsell 100-Hue Test. The total error score was derived by counting the number of caps misplaced.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: total error score
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
total error score
  Right eye | 0.1 (1.98) | -0.4 (2.37)
  Left eye | -0.2 (1.70) | -0.5 (1.99)
Statistical Analysis 1: Comparison: Active vs Placebo; The sample size had enough power to detect any meaningful difference between treatment groups in the right eye; Test type: Superiority or Other; p = 0.8216, ANCOVA; LS mean difference = 0.076, 95% CI 2-sided [-0.592 to 0.744], Standard Error of Mean 0.335
Statistical Analysis 2: Comparison: Active vs Placebo; The sample size had adequate power to detect a meaningful difference between treatment groups in the left eye; Test type: Superiority or Other; p = 0.324, ANCOVA; LS means difference = 0.257, 95% CI 2-sided [-0.258 to 0.771], Standard Error of Mean 0.258

2. Primary Outcome: Change From Baseline in Visual Acuity 1 Hour Post Dosing
Description: Visual acuity was measured using the Logarithm of the Minimum Angle Resolution (LogMAR) chart. The LogMAR value of the best line read was noted and the number of letters read in the next row was multiplied by 0.02, then subtracted from the LogMAR value of the best line completely read.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
LogMar
  Right Eye | -0.014 (0.0641) | -0.023 (0.0694)
  Left Eye | -0.042 (0.0809) | -0.011 (0.0836)
Statistical Analysis 1: Comparison: Active vs Placebo; The sample size provided enough power to detect any meaningful difference between the two treatment groups in the right eye; Test type: Superiority or Other; p = 0.7864, ANCOVA; LS means difference = 0.004, 95% CI 2-sided [-0.024 to 0.031], Standard Error of Mean 0.014
Statistical Analysis 2: Comparison: Active vs Placebo; The sample size provided enough power to detect any meaningful difference between the two treatment groups in the left eye; Test type: Superiority or Other; p = 0.1953, ANCOVA; LS Means difference = -0.022, 95% CI 2-sided [-0.056 to 0.012], Standard Error of Mean 0.017

3. Primary Outcome: Change From Baseline in Pupil Dilation 1 Hour Post Dosing
Description: Pupil dilation was measured using the Neuroptics Model VIP 200 pupillometer under standard lighting conditions.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
millimeter
  Right eye | -0.14 (0.280) | 0.02 (0.270)
  Left eye | -0.19 (0.264) | -0.10 (0.285)
Statistical Analysis 1: Comparison: Active vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0101, ANCOVA; LS means difference = -0.160, 95% CI 2-sided [-0.280 to -0.039], Standard Error of Mean 0.061
Statistical Analysis 2: Comparison: Active vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1583, ANCOVA; LS means difference = -0.087, 95% CI 2-sided [-0.209 to 0.035], Standard Error of Mean 0.061

4. Primary Outcome: Change From Baseline in Intraocular Pressure 1 Hour Post Dosing
Description: Intraocular Pressure was measured using the Goldman applanation tonometry
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
mm Hg
  Right eye | 0.03 (1.761) | 0.29 (1.609)
  Left eye | 0.36 (1.860) | -0.26 (1.335)
Statistical Analysis 1: Comparison: Active vs Placebo; The sample size should provide approximately 90% power to detect a 1.6 mmHg difference in the mean change in Intraocular Pressure between the two treatment groups in the right eye; Test type: Superiority or Other; p = 0.9324, ANCOVA; LS means difference = -0.031, 95% CI 2-sided [-0.746 to 0.685], Standard Error of Mean 0.359
Statistical Analysis 2: Comparison: Active vs Placebo; The sample size should provide approximately 90% power to detect a 1.6 mmHg difference in the mean change in intraocular pressure between the two treatment groups in the left eye; Test type: Superiority or Other; p = 0.0343, ANCOVA; LS means difference = 0.751, 95% CI 2-sided [0.057 to 1.44], Standard Error of Mean 0.348

5. Secondary Outcome: Change From Baseline in Visual Acuity 24 Hours Post Dosing
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
LogMar
  Right eye | -0.012 (0.0682) | -0.035 (0.0920)
  Left eye | -0.027 (0.1042) | -0.020 (0.0908)
Statistical Analysis 1: Comparison: Active vs Placebo; The sample size had enough power to detect any meaningful difference between treatment groups in the right eye; Test type: Superiority or Other; p = 0.3139, ANCOVA; LS Means difference = 0.017, 95% CI 2-sided [-0.017 to 0.051], Standard Error of Mean 0.017
Statistical Analysis 2: Comparison: Active vs Placebo; The sample size had enough power to detect any meaningful difference between treatment groups in the left eye; Test type: Superiority or Other; p = 0.9334, ANCOVA; LS means difference = -0.002, 95% CI 2-sided [-0.045 to 0.042], Standard Error of Mean 0.022

6. Secondary Outcome: Change From Baseline in Pupil Dilation 24 Hour Post Dosing
Time Frame: 24 hour
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
mm
  Right eye | 0.0 (0.238) | -0.02 (0.249)
  Left eye | -0.06 (0.223) | -0.07 (0.289)
Statistical Analysis 1: Comparison: Active vs Placebo; The sample size had enough power to detect any meaningful difference between treatment groups in the right eye; Test type: Superiority or Other; p = 0.7723, ANCOVA; LS means difference = 0.016, 95% CI 2-sided [-0.093 to 0.125], Standard Error of Mean 0.055
Statistical Analysis 2: Comparison: Active vs Placebo; The sample size had enough power to detect any meaningful difference between treatment groups in the left eye; Test type: Superiority or Other; p = 0.9107, ANCOVA; LS means difference = 0.007, 95% CI 2-sided [-0.109 to 0.122], Standard Error of Mean 0.058

7. Secondary Outcome: Change From Baseline in Color Vision Discrimination 24 Hour Post Dosing
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: total error score
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
total error score
  Right eye | -0.1 (1.66) | -0.4 (2.49)
  Left eye | -0.2 (1.69) | -0.1 (2.14)
Statistical Analysis 1: Comparison: Active vs Placebo; The sample size had enough power to detect any meaningful difference between treatment groups in the right eye; Test type: Superiority or Other; p = 0.7787, ANCOVA; LS Means difference = -0.078, 95% CI 2-sided [-0.632 to 0.475], Standard Error of Mean 0.278
Statistical Analysis 2: Comparison: Active vs Placebo; The sample size had enough power to detect any meaningful difference between treatment groups in the left eye; Test type: Superiority or Other; p = 0.6013, ANCOVA; LS means difference = -0.180, 95% CI 2-sided [-0.865 to 0.504], Standard Error of Mean 0.344

8. Secondary Outcome: Change From Baseline in Intraocular Pressure 24 Hour Post Dosing
Description: Intraocular pressure was measuring using the Goldman applanation tonometry
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Active | Placebo
Number analyzed (Participants) | 40 | 40
mm Hg
  Right eye | -0.10 (2.176) | 0.03 (1.423)
  Left eye | 0.03 (1.694) | -0.09 (1.339)
Statistical Analysis 1: Comparison: Active vs Placebo; The sample size should provide approximately 90% power to detect a 1.6 mmHg difference in the mean change in IOP between the two treatment groups in the right eye; Test type: Superiority or Other; p = 0.8209, ANCOVA; LS means difference = 0.091, 95% CI 2-sided [-0.705 to 0.887], Standard Error of Mean 0.400
Statistical Analysis 2: Comparison: Active vs Placebo; The sample size should provide approximately 90% power to detect a 1.6 mmHg difference in the mean change in IOP between the two treatment groups in the left eye; Test type: Superiority or Other; p = 0.4931, ANCOVA; LS means difference = 0.227, 95% CI 2-sided [-0.430 to 0.884], Standard Error of Mean 0.330

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 16/40 | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=40) | Placebo (N=40)
abdomonial pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
feeling hot (General disorders) | 2 (2) | 0 (0)
alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
blood urine present (Investigations) | 1 (1) | 0 (0)
protein urine present (Investigations) | 1 (1) | 0 (0)
red blood cells urine (Investigations) | 2 (2) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 10 (10) | 1 (1)
libido increased (Psychiatric disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
flushing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days